CLINICAL TRIAL: NCT00173121
Title: Environmental Enterovirus Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700414
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-04

CONDITIONS: Transmission Condition
Keywords: enterovirus, environment, aerosol, air
MeSH Terms: conditions — Enterovirus Infections

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
From last decades, because of lacking the powerful quantitative methods, such as real-time qPCR, there is no environmental monitoring data about enterovirus transmission. If the major transmission routes and risk factor are still not clear, it will be very hard for making the prevention and control strategies. Today, the most popular prevention suggestion for children is keeping them away from crowded public places during the peak contagious season, because enteroviruses are easily transmitted through aerosols over a distance of meters, and even between separated rooms (Chang et al., 2004). However, adults may as easily be infected, but don』t have any disease symptoms or carry the virus home. Another recommendation is washing hands to avoid contact of hands or anything else with the mouth and nose, as it is through contact of viruses with the mucosal membranes in the mouth and nasal passages that infection occurs. However, these actions did not be great helpful for preventing enterovirus infection and spread. Understanding and disrupting the major transmission pass way of enterovirus could be more effective than just keeping personal hygiene. Therefore, an applicable environmental monitoring program is needed for understanding the transmission routes and risk factor of enterovirus infection. In this study, we will monitor enteroviruses in hospital, household and kindergarten. For the environmental monitoring of enteroviruses, we will apply traditional plaque assay, real-time quantitative PCR and combine with questionnaire-based interviews to understand the infectious types and concentration of enterovirus from indoor air, surface and water for recognizing the transmission routes of enterovirus and the relationships between virus concentration and the symptoms of the cases.

DETAILED DESCRIPTION:
Environmental Monitoring Program for Enterovirus (1) Case Collection. The studies cases include patients who were suspected of having enterovirus illnesses, such as HFMD and herpangina. Institutional review board approval was obtained from the Hospital for this study and informed consent was obtained from all patients or their parents. (2) Questionnaire. questionnaire based interviews were used to collect information about the family members, including demographic data, the number of bedrooms in the house, amount of contact time with the patient, presence and pattern of current or recent signs and symptoms. (3) Patient and culture samples. Laboratory evidence of enterovirus infection was defined as the isolation of enterovirus from a throat , and rectal swab sample. (4) Environmental Sampling. (a) Air sampling. For the filter/real-time qPCR assay, the air in each ward was filtered through a 37-mm-diameter Nuclepore filter (Costar, Cambridge, MA), which is a track-etched polycarbonate filter consisting of a polycarbonate membrane with straight-through pores of uniform size (0.4 μm). The filters were supported by cellulose pads and loaded into open-face three-piece plastic cassettes. The pump and filter apparatus were placed within 1 m from the patient's bed on an adjacent nightstand. (b) Surface sampling Regarding surface sampling, surfaces of environment and equipment were sampled with moistened sterile cotton swabs.

ELIGIBILITY:
Inclusion Criteria:

* any case of enterovirus infection

Exclusion Criteria:

* not enterovirus infection cases

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2005-05; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Luan-Yin Chang Chang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hsopital, Taipei, Taipei, Taiwan